CLINICAL TRIAL: NCT03402568
Title: Circulating Metabolites Associated With Alcohol Intake in the European Prospective Investigation Into Cancer and Nutrition Cohort
Brief Title: Alcohol Consumption and Circulating Metabolites
Status: Completed | Type: Observational
Sponsor: International Agency for Research on Cancer (Other)
Collaborators: Maastricht University (Other); Imperial College London (Other); Danish Cancer Society (Other); University of Aarhus (Other); Centre for Research in Epidemiology and Population Health (CESP) (Other); Gustave Roussy, Cancer Campus, Grand Paris (Other); German Cancer Research Center (Other); German Institute of Human Nutrition (Other); Hellenic Health Foundation (Other); Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); ISPO Cancer Prevention and Research Institute (Unknown); Federico II University (Other); HuGeF Foundation (Unknown); Azienda Sanitaria Provinciale Ragusa (Other); University of Tromso (Other); Institut Català d'Oncologia (Other); Ministry of Health - Government of the Principality of Asturias (Other Government); Andalusian School of Public Health (Other Government); Universidad de Murcia (Other); Instituto de Salud Pública Gobierno de Navarra (Unknown); Subdirección de Salud Pública de Gipuzkoa (Unknown); Skane University Hospital (Other); Umeå University (Other); MORGEN-EPIC, Bilthoven (Unknown); Prospect-EPIC, Utrecht (Unknown); University of Oxford (Other); University of Cambridge (Other)
Responsible Party: Sponsor
Other Study IDs: PP201712-35
Record Dates: First submitted 2018-01-10; First posted 2018-01-18 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: No Condition, Focus: Metabolites of Alcohol Consumption
Keywords: alcohol; targeted metabolomics; lipid metabolites; amino acids; acylcarnitines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum and citrate plasma blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Alcohol consumption is a risk factor for numerous health conditions and an important cause of death. Identifying metabolites associated with alcohol consumption may provide insights into the metabolic pathways through which alcohol may affect human health. The objective of this study is to investigate associations of alcohol consumption with circulating concentrations of 123 metabolites including amino acids, acylcarnitines, hexoses, biogenic amines, phosphatidylcholines, and sphingomyelins. For this purpose, the investigators use data from the European Prospective Investigation into Cancer and Nutrition (EPIC) study and applied a discovery and replication approach.

DETAILED DESCRIPTION:
This study used data from 2,974 control participants from four case-control studies on colorectal (n=491), hepatobiliary (n=327), kidney (n=635), and prostate cancer (n=1,521) nested in the EPIC cohort, for which targeted metabolomics data had been acquired. Alcohol consumption at recruitment was self-reported through dietary questionnaires. Metabolite concentrations were measured by tandem mass spectrometry using the BIOCRATES AbsoluteIDQTM p180 kit. Data were randomly divided into discovery (2/3) and replication (1/3) sets. Multivariable linear regression models were used to evaluate confounder-adjusted associations of ln-transformed alcohol consumption with Z-standardized ln-transformed residual metabolite concentrations. Metabolites significantly related to alcohol intake in the discovery set (FDR q-value<0.05) were further tested in the replication set (Bonferroni-corrected p-value<0.05). Of the 72 metabolites significantly related to alcohol intake in the discovery set, 34 metabolites were also significant in the replication analysis, including three acylcarnitines, the amino acid citrulline, four lysophosphatidylcholines, 13 diacylphosphatidylcholines, seven acyl-alkylphosphatidylcholines, and six sphingomyelins. Associations with acylcarnitines and phosphatidylcholines were generally positive, while mostly inverse associations were observed with citrulline and sphingomyelins.

This study adds novel knowledge regarding circulating metabolites associated with alcohol consumption, and provides leads for further studies into the underlying biological mechanisms. A better understanding of metabolic pathways affected by alcohol consumption may contribute to the development of mechanism-tailored intervention strategies to prevent and treat alcohol-related conditions. Furthermore, it may help to identify biomarkers of alcohol consumption facilitating early preventive strategies in individuals at-risk for developing alcohol-related morbidities.

ELIGIBILITY:
Inclusion Criteria (for EPIC):

* Aged 30-70
* Healthy volunteers residing within defined geographical areas (where study centers are located). Different settings by centre; mostly general population with some exceptions: women of a health insurance company for teachers and school workers (France), women attending breast cancer screening (Utrecht-The Netherlands, and Florence-Italy), mainly blood donors (most centers in Italy and Spain) and a cohort consisting predominantly of vegetarians (the 'health-conscious' group in Oxford, UK).

Exclusion criteria (for this study):

* Individuals without metabolomics data
* Individuals without data on alcohol consumption at recruitment

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Over 520,000 healthy men and women aged 25-85 were enrolled between 1992 and 2000 across 23 EPIC centres in 10 European countries including Denmark, France, Germany, Greece, Italy, the Netherlands, Norway, Spain, Sweden, and the United Kingdom.
  This study used data from 2,974 control participants from four case-control studies on colorectal (n=491), hepatobiliary (n=327), kidney (n=635), and prostate cancer (n=1,521) nested in the EPIC cohort, for which targeted metabolomics data had been acquired.
Sampling Method: Probability Sample
Enrollment: 2974 (Actual)
Dates: Start 2012-10-24 (Actual); Primary Completion 2016-10-26 (Actual); Study Completion 2016-10-26 (Actual)

PRIMARY OUTCOMES:
Circulating metabolite concentrations | Laboratory analyses performed between Oct 2012-Oct 2016
  Blood concentrations of 123 metabolites including amino acids, acylcarnitines, hexoses, biogenic amines, phosphatidylcholines, and sphingomyelins (BIOCRATES AbsoluteIDQTM p180 kit).

IPD SHARING:
Plan to Share IPD: Undecided
Undecided.